CLINICAL TRIAL: NCT06033508
Title: Effects of Whole-body Vibration Therapy on Type 2 Diabetic Patients with and Without Polyneuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, GULIN FINDIKOGLU, Assoc Prof Dr, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-60116787-020-338517
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes; Diabetic Peripheral Neuropathy; Exercise
Keywords: Type 2 diabetes mellitus; Diabetic Peripheral Neuropathy; whole body vibration; inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Inflammation | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- T2DM with neuropathy + WBV (Active Comparator): Patients with type 2 Diabetes mellitus with neuropathy who will be trained by whole body vibration
  Interventions: Other: exercise with whole body vibration device
- T2DM without neuropathy + WBV (Active Comparator): Patients with type 2 Diabetes mellitus without neuropathy who will be trained by whole body vibration
  Interventions: Other: exercise with whole body vibration device
- T2DM without neuropathy + land exercise (Placebo Comparator): Patients with type 2 Diabetes mellitus without neuropathy who will be trained on land
  Interventions: Other: placebo exercise

INTERVENTIONS:
Other: exercise with whole body vibration device — exercise with whole body vibration device
  Arms: T2DM with neuropathy + WBV; T2DM without neuropathy + WBV
Other: placebo exercise — exercise without vibration on land
  Arms: T2DM without neuropathy + land exercise

SUMMARY:
The aim of this study is to show how whole body vibration training practiced for 12 weeks affects the levels of inflammatory biomarkers such as C reactive protein (CRP) and, interleukin-6 (IL-6), in Type 2 diabetic patients (T2DM) with and without peripheral neuropathy.

DETAILED DESCRIPTION:
Volunteers with type 2 diabetes mellitus with and without peripheric neuropathy will be evaluated in terms of any contra-indication that will restrain them from making exercise with whole body vibration device. 60 male or female volunteers who are suitable in terms of inclusion/exclusion criteria will be invited for the study. Volunteers will be randomly distributed to one of the 3 groups. Each group will contain 20 participants. 1st group will include type 2 diabetic patients with peripheric neuropathy and 2nd and 3rd groups will include type 2 diabetic patients without neuropathy. Patients in group 1 and 2 will make static isometric exercises on vibration platform whereas patients in group 3 will make the same exercises on land in the hospital setting. Participants will be requested to complete 3 months of exercise. They will be evaluated before and at the end of the 3 months of exercise with physical measures such as waist and hip circumference, 6-minute walk test, body composition measured by bioimpedance, muscle thickness, and blood tests to measure inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must stand and walk o without using an assistive device.
2. Participants must have a weight of less than 120 kg.

Exclusion Criteria:

1. T2DM patients with advanced cardiovascular, renal, hepatic disease
2. T2DM patients with diabetic retinopathy or nephropathy
3. T2DM patients with untreated hypertension, rhythm disorders, and those who have undergone bypass surgery
4. T2DM patients with ischemic changes in the resting ECG
5. T2DM patients with untreated hypoglycemia or orthostatic hypotension
6. T2DM patients who are unable to walk independently, or use of canes, crutches or wheelchairs
7. T2DM patients who have open ulcers or wounds on load-bearing surfaces
8. T2DM patients with inflammatory rheumatic diseases such as rheumatoid arthritis
9. T2DM patients with active infectious disease
10. T2DM patients with high risk of thrombosis, those with deep vein thrombosis
11. T2DM patients who carry a pacemaker, prosthesis, intrauterine device or metal implant,
12. T2DM patients with a history of cancer
13. T2DM patients with severe migraine, epilepsy, stroke or other neurological disorders, those who have undergone brain surgery
14. T2DM patients with non-diabetic neuropathy due to reasons such as HIV, AIDS, alcohol, uremia
15. T2DM patients with cognitive impairment
16. T2DM patients who are on psychotropic or neurotoxic therapy
17. T2DM patients with advanced balance problems
18. T2DM patients who are pregnant or breastfeeding mothers
19. T2DM patients who are organ transplant recipients
20. T2DM patients with hernia
21. T2DM patients with kidney or bladder stones
22. T2DM patients who are exposed to mechanical vibration due to their job

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
6 min walk test | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GULIN FINDIKOGLU, Assoc Prof, Principal Investigator — Pamukkale University, Medical Faculty, PMR Department
Locations (1):
- Pamukkale University, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No